CLINICAL TRIAL: NCT00127010
Title: Blinded, Randomized Study to Evaluate the Immunogenicity and Safety of GlaxoSmithKline Biologicals' Measles-mumps-rubella-varicella Candidate Vaccine Given to Healthy Children During the Second Year of Life
Brief Title: Immunogenicity and Safety of a Combined Vaccine to Prevent Measles, Mumps, Rubella and Chickenpox Diseases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 103388
Record Dates: First submitted 2005-08-04; First posted 2005-08-05 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Measles; Rubella; Mumps; Varicella
Keywords: Prophylaxis measles, mumps, rubella and chickenpox
MeSH Terms: conditions — Measles; Rubella; Mumps; Chickenpox | interventions — Vaccines, Attenuated

INTERVENTIONS:
Biological: Measles, Mumps, Rubella and Chickenpox (live vaccine)
  Other Names: Measles; Mumps; Rubella and Chickenpox (live vaccine)

SUMMARY:
This is a study to evaluate the immunogenicity and safety of GlaxoSmithKline (GSK) Biologicals combined measles-mumps-rubella varicella candidate vaccine given to healthy children in their second year of life.

DETAILED DESCRIPTION:
This study included an active control group who received the licensed Priorix (measles, mumps, rubella [MMR] vaccine).

ELIGIBILITY:
Inclusion Criteria:

* A male or female subject between 11-13 months of age (i.e. from 11 month birthday until the day before the 14 month birthday) at the time of the first vaccination.

Exclusion Criteria:

* History of previous measles, mumps, rubella and/or varicella vaccination or disease, or known exposure to any of these diseases within 30 days prior to the start of the trial
* Planned administration of a vaccine not foreseen by the study protocol from 30 days prior to each vaccination until 42-56 days after each vaccination

Ages: 11 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2005-11; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Antibody levels after vaccination

SECONDARY OUTCOMES:
Safety of the study vaccines

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (47):
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
- Germany (44):
  - GSK Investigational Site, Bad Saulgau, Baden-Wurttemberg
  - GSK Investigational Site, Bönnigheim, Baden-Wurttemberg
  - GSK Investigational Site, Ehingen, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Kirchzarten, Baden-Wurttemberg
  - GSK Investigational Site, Ludwigsburg, Baden-Wurttemberg
  - GSK Investigational Site, Marbach, Baden-Wurttemberg
  - GSK Investigational Site, Oberkirch, Baden-Wurttemberg
  - GSK Investigational Site, Offenburg, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tauberbischofsheim, Baden-Wurttemberg
  - GSK Investigational Site, Tettnang, Baden-Wurttemberg
  - GSK Investigational Site, Bindlach, Bavaria
  - GSK Investigational Site, Cham, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Weilheim, Bavaria
  - GSK Investigational Site, Werneck, Bavaria
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Niedernhausen, Hesse
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Espelkamp, North Rhine-Westphalia
  - GSK Investigational Site, Herford, North Rhine-Westphalia
  - GSK Investigational Site, Hille, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Minden, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Porta Westfalica, North Rhine-Westphalia
  - GSK Investigational Site, Viersen, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Brunsbüttel, Schleswig-Holstein
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Glücksburg, Schleswig-Holstein
  - GSK Investigational Site, Husum, Schleswig-Holstein
  - GSK Investigational Site, Neumünster, Schleswig-Holstein
  - GSK Investigational Site, Neuhaus am Rennweg, Thuringia
- GSK Investigational Site, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 103388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 103388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 103388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 103388 are summarised with followup study 104690 on the GSK Clinical Study Register.
- Available data/document: Informed Consent Form: 103388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 103388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register